CLINICAL TRIAL: NCT06952933
Title: Psychological Trauma, Post-Traumatic Stress Disorder, and Resilience in Adults With Congenital Heart Disease
Acronym: PTSD in ACHD
Status: Not yet recruiting | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Adult Congenital Heart Association (Unknown)
Responsible Party: Principal Investigator, David J. Harrison, Assistant Professor, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02002388
Record Dates: First submitted 2025-01-08; First posted 2025-05-01 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Adult Congenital Heart Disease; Congenital Heart Disease; PTSD
Keywords: adult congenital heart disease; achd; congenital heart disease; pediatric cardiology; ptsd; post-traumatic stress disorder; resilience
MeSH Terms: conditions — Heart Defects, Congenital; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Overall cohort: Adults age >= 18-years with a diagnosis of congenital heart disease.
  Congenital heart disease will be defined by previously published classification including those listed in the American Heart Association/ American College of Cardiology guidelines for the care of adults with congenital heart disease.
  Interventions: Behavioral: Other

INTERVENTIONS:
Behavioral: Other — Surveys will be distributed for data collection. A subset of patients will participate in diagnostic clinician interviews. No interventions will be tested.
  Other Names: Assessment of PTSD symptoms and resilience

SUMMARY:
The purpose of this study, entitled "Psychological trauma, post-traumatic stress disorder, and resilience in adults with congenital heart disease in a large population sample", is to evaluate for exposures during a lifetime with congenital heart disease that may be associated with higher likelihood of developing PTSD.

Primary aim:

- Identify individual patient characteristics (medical, psychosocial, socioeconomic, etc.) that are associated with a diagnosis of PTSD.

Secondary aims:

* Calculate the prevalence of those meeting PTSD criteria in the ACHD population using the "gold standard" diagnostic clinician interview, while using the same data to validate a PTSD screening self-report survey in the ACHD population.
* Determine the role of resilience in ACHD patients using a validated screening survey to assess its protective role toward PTSD.

Hypotheses:

* There are certain exposures (e.g. post-surgical pain, ICU delirium, bullying due to CHD) that are associated with a higher incidence and odds of meeting PTSD criteria.
* "Gold standard" diagnostic interviews will most accurately estimate the prevalence of PTSD in ACHD which has been overestimated on prior screening-based studies, although the scope of the problem is still great.
* Patients with a higher resilience score will show an association with a lower risk of PTSD.

DETAILED DESCRIPTION:
The purpose of this study, entitled "Psychological trauma, post-traumatic stress disorder, and resilience in adults with congenital heart disease in a large population sample", is to evaluate for exposures during a lifetime with congenital heart disease that may be associated with higher likelihood of developing PTSD.

This study will use the existing registry for the Congenital Heart Initiative (CHI), which contains over 4,000 ACHD patients who have opted in to receive surveys from this research team. The CHI was launched in late 2020, and full information can be found at [clinicaltrials.gov ID: NCT05185232]. For this PTSD and resilience arm of the study, an email invitation will be sent to all CHI members, who can opt in to complete surveys assessing psychological trauma as a consequence of one's heart disease.

The first stage will be a distribution of approximately two surveys. The first survey is called the Post-traumatic Stress Disorder Checklist for the DSM-5 (PCL-5), a 20-item screening tool with a score ranging from 0 (no symptoms) to 80 (highest symptoms). As a screener, this survey does not diagnose PTSD, but identifies those who are experiencing significant symptoms. Because of the sensitive nature of this topic, all survey items are optional and there is no penalty for not finishing the survey.

The next survey will study resilience, most likely using the Connor-Davidson Resilience Scale, which has been tested in other ACHD studies. Resilience is defined as a person's ability to withstand and recover from stressful life experiences. Studying resilience will serve as an ideal balancing measure to the study of PTSD.

The final stage of this study will be in-person diagnostic interviews. Trained psychology research assistants will help administer the Clinician Administered PTSD Diagnostic Interview (CAPS-5) via video conference. Recruitment for this phase will include a subset of respondents who are invited from those who completed the PCL-5 to participate in the CAPS-5 if they choose to do so. This will include all ranges of scores on the PCL-5, representing those who screen positive and negative using the PCL-5. The CAPS-5 is considered the gold standard for PTSD diagnosis, and can provide valuable validation information for the PCL-5 in this population. At the conclusion of the interview, the study team may discuss resilience-building strategies as a qualitative assessment.

Overall, the investigators aim to estimate the prevalence of psychological trauma and PTSD in the ACHD population, as well as learning strategies to build resilience. This study will also aim to validate the screening tools for PTSD and resilience, so they may be implemented in the outpatient setting. The study team will assess for conditions that are most associated with PTSD and resilience, to help identify patients who may be at higher risk based on their illness course. Stressful experiences such as surgeries, arrhythmias, ICU admissions, and general anxiety about one's heart may be unavoidable at times. By understanding what drives a patient's illness experience, clinicians can plan for interventions to reduce trauma and build resilience.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease diagnosis, age >= 18 years
* Enrolled in CHI registry
* English proficiency for survey completion
* Access to an internet connection. Can be via computer or handheld device.

Exclusion Criteria:

* Any who opt out
* Age < 18 years
* No diagnosis of congenital heart disease
* Not enrolled in CHI registry/unable to access Internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult with a congenital heart disease diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
PTSD checklist for DSM-5 (PCL-5) | One-time survey. Distribute to patients during months ~1-2.
  A 20-item survey of the five domains of PTSD as described by the DSM-5. Each item is on a five-point Likert scale describing severity of symptoms (bothered by symptoms "not at all" to "extremely"). Each item is graded 0 to 4, for a total PCL-5 score ranging from 0 to 80. Historical studies have recommended a cutoff for PTSD-positive around 31 to 33. This study will attempt to validate the proper cutoff in the ACHD population using the diagnostic interview.

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale Diagnostic Interview (CAPS-5) | One-time interview during study months 4 to 12
  For a subset of patients: The CAPS-5 scoring system ranges from 0 to 80, with measures for symptom severity and frequency for each of the PTSD symptom clusters as defined by the DSM-5. Questioning and scoring will be performed by trained facilitators who will conduct the diagnostic interview via video conference. A higher score indicates more severe symptoms, while the presence of symptoms for each symptom cluster is required to confirm a diagnosis of PTSD.
Connor-Davidson Resilience Scale (CD-RISC) | One-time survey. Distribute to patients during months ~1-2.
  A 10-item survey of statements that are associated with resilience. Respondents will indicate their level of agreement on a 5-point Likert scale (range 0 to 4), for a total score of 0 to 40. A higher score indicates a higher level of resilience.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
This study is not a clinical trial and does not have an intervention group. Some data collected will be on sensitive topics. No current plan to share data with other researchers.

REFERENCES:
- [Background] Webb G, Landzberg MJ, Daniels CJ. Specialized adult congenital heart care saves lives. Circulation. 2014 May 6;129(18):1795-6. doi: 10.1161/CIRCULATIONAHA.114.009049. Epub 2014 Mar 3. No abstract available. PMID 24589850
- [Background] Steiner JM, Nassans K, Brumback L, Stout KK, Longenecker CT, Yi-Frazier JP, Curtis JR, Rosenberg AR. Key Psychosocial Health Outcomes and Association With Resilience Among Patients With Adult Congenital Heart Disease. JACC Adv. 2024 May;3(5):100917. doi: 10.1016/j.jacadv.2024.100917. Epub 2024 Mar 28. PMID 38846320
- [Background] Phillippi R, Leezer S, Messmer M, Hile D, John AS. Patient Engagement in Research: Considerations in Creating a Registry for Adults with Congenital Heart Disease. Curr Cardiol Rep. 2024 Jan;26(1):15-21. doi: 10.1007/s11886-023-02013-2. Epub 2023 Dec 22. PMID 38133788
- [Background] Harrison DJ, Kay J, Jacobsen RM, Londono-Obregon C, Yeung E, Kelly SL, Poteet A, Levek C, Landzberg MJ, Wallrich M, Khanna A. The burden of psychological trauma and post-traumatic stress disorder among adults with congenital heart disease: PTSD in ACHD. Am J Cardiol. 2024 May 15;219:9-16. doi: 10.1016/j.amjcard.2024.03.007. Epub 2024 Mar 6. PMID 38458583
- See also: Congenital Heart Initiative enrollment page — https://www.achaheart.org/your-heart/programs/research/join-the-congenital-heart-initiative/